CLINICAL TRIAL: NCT06016465
Title: Does Nerve Block Plus Oral Dexamethasone Reduce Recurrence of Headache Within 72 Hours Better Than Nerve Block Alone?
Brief Title: Does Nerve Block + Oral Dexamethasone Reduce Recurrence of Headache Within 72 Hrs?
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Edward Michelson, MD, Professor and Chair Dept of Emergency Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E23081
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: migraine headache; peripheral nerve block; dexamethasone; steroid treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 for study drug vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study drug pills (dexamethasone or placebo) will be placed in identical colored capsules and then into numbered packets. Only pharmacist will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): single oral dose of dexamethasone (8mg)
  Interventions: Drug: Dexamethasone Oral
- Placebo (Placebo Comparator): Single oral dose of placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone Oral — Two 4mg pills
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Placebo — 2 placebo pills
  Other Names: Dextrose methyl cellulose
  Arms: Placebo

SUMMARY:
For some patients who come to the emergency department for treatment of a migraine headache, peripheral headache nerve blocks (PHNB) have proven to be an efficient and effective treatment for headache relief. Previous studies have demonstrated that adding steroids as an adjunct treatment to standard migraine treatment can reduce recurrence of headaches in the subsequent few days.

DETAILED DESCRIPTION:
Previous studies have provided evidence that administering steroids in addition to standard migraine headache treatment in the emergency department may reduce the recurrence of the headache within 24-72 hours. The standard migraine treatments in previous studies have been varied and include 5-HT receptor agonists, dopamine antagonists, dihydroergotamine, NSAIDS, and opioid analgesics. The steroids added to the standard treatment have been prednisone and dexamethasone (both IV and oral).

This is the first study to examine the combination of peripheral nerve block as the primary treatment of migraine followed by oral dexamethasone to prevent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Meet ICHD-3 Migraine Headache Criteria
* Had a minimum 5-point reduction in headache intensity after nerve block(s) or post- block pain score of 0 to 2
* Nerve block performed with bupivacaine 0.5%

Exclusion Criteria:

* Head trauma
* Suspicion of secondary headache (i.e. stroke, known tumor, glaucoma)
* Headache in the setting of viral syndrome
* Chronically on steroids
* Known allergy to dexamethasone
* Unable to reach the patient by phone or text for follow-up
* Gestational diabetes or other uncontrolled diabetes
* Known to be immunocompromised

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of headache | 72-96 hours post treatment
  Subjects will be contacted 72 hrs post treatment to determine if migraine headache has recurred

SECONDARY OUTCOMES:
Early recurrence headache and timing | 72-96hrs post treatment
  HA severity, location, time since enrollment enrollment,medications
side effects of dexamethasone identified if any | 72-96 hrs post treatment
  elevation in glucose level, other symptoms associated with corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Susan Watts, PhD., Study Director — Texas Tech University Health Sciences Center, Department of Emergency Medicine
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No